CLINICAL TRIAL: NCT06785467
Title: eDoula: The Feasibility and Acceptability of Mobile Application in Pregnancy, Labor, and Birth Support
Brief Title: eDoula Feasibility and Acceptability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Fei Cai, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB 27596
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Related
Keywords: Labor; Birth

STUDY DESIGN:
Intervention Model Description: Control group will receive routine care and will be recruited postpartum to respond to a survey on their labor and satisfaction outcomes. Once control group recruitment is complete, intervention recruitment will begin. Intervention arm participants will gain access to the eDoula app during pregnancy.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): These participants will receive routine pregnancy and delivery care.
- eDoula Intervention (Experimental): These participants will have access to the eDoula app during pregnancy.
  Interventions: Other: eDoula App

INTERVENTIONS:
Other: eDoula App — eDoula is an app that will give patients reading material and videos to watch based on their due date. It also provides helpful postpartum device.
  Arms: eDoula Intervention

SUMMARY:
eDoula is an app that will give patients reading material and videos to watch based on their due date. It also provides helpful postpartum guidance. First, patients without access to the app will be recruited and surveyed on their labor and satisfaction outcomes. Then, recruitment will begin for the intervention arm of the study. Participants will be recruited to use the app and complete a survey during the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* Singleton pregnancy
* English speaking
* Own a smart phone or other device capable of downloading and running the eDoula app
* Delivered at 36 weeks 0 days gestation or later
* Able to labor

Exclusion Criteria:

* Planned cesarean delivery
* Pregnancy complications including placenta accreta spectrum, vasa previa, intrauterine fetal demise, or known major fetal anomaly
* Delivery planned at a location other than Oregon Health and Science University

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with eDoula app | Measured in the 7 days following delivery
  Participant-reported satisfaction with the eDoula app using a 3-question Likert scale. Scores can have a value from 3 to 15, with a higher score indicating greater satisfaction.
eDoula App Use | Recruitment (19-28 weeks gestation) to delivery
  The number of days during pregnancy that the eDoula app was used

SECONDARY OUTCOMES:
Labor Agentry Scale-10 (LAS-10) | Measured in the 7 days following delivery
  Instrument measuring patient control during childbirth. Scores can have a value from 10 to 70, with a higher score indicating a better outcome.
Birth Satisfaction Scale-Revised (BSS-R) | Measured in the 7 days following delivery
  Instrument measuring patient satisfaction with the birth experience. Scores can have a value from 0 to 40, with higher scores representing greater birth satisfaction.
Edinburgh Postnatal Depression Scale (EPDS) | Measured in the 7 days following delivery
  Instrument measuring postnatal depression symptoms following delivery. Scores can have a falue from 0 to 30, with higher scores representing more symptoms of postnatal depression.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Cai, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No